CLINICAL TRIAL: NCT04102592
Title: IGHID 11829 - Getting Malaria "Off the Back" of Women and Children in Western Uganda
Brief Title: Getting Malaria "Off the Back" of Women and Children in Western Uganda
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Conservation, Food, and Health Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 18-1819; IGHID 11829 (Other: University of North Carolina at Chapel Hill)
Record Dates: First submitted 2019-09-23; First posted 2019-09-25 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-02

CONDITIONS: Malaria
Keywords: Malaria; P. Falciparum; Permethrin; Rapid diagnostic test
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to control (25) or intervention group (25)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants in this arm receive Lesu (baby wrap) treated with 0.5% permethrin
  Interventions: Other: Permethrin-treated Lesu (baby wrap)
- Control Group (Placebo Comparator): Participants in this arm receive Lesu (baby wrap) soaked with water only to mimic re-treatment and mask allotment
  Interventions: Other: Untreated Lesu (baby wrap)

INTERVENTIONS:
Other: Permethrin-treated Lesu (baby wrap) — 0.5% permethrin application
  Arms: Intervention Group
Other: Untreated Lesu (baby wrap) — Matching untreated lesu
  Other Names: Placebo
  Arms: Control Group

SUMMARY:
This is a two-phase, mixed-methods pilot study of insecticide-treated lesus to reduce the incidence of P. falciparum malaria among infants in a rural area of western Uganda. Participants will be recruited from four villages immediately adjacent to the Bugoye Level III Health Centre (Bugoye, Kanyanamigho, Izinga, Rwakingi 1a) in the Kasese District of western Uganda.

The purpose of the study is to assess the feasibility and tolerability of using insecticide-treated lesus to reduce the incidence of P. falciparum malaria infection among infants.

DETAILED DESCRIPTION:
This is a two-phase, mixed-methods pilot study of insecticide-treated lesus to reduce the incidence of P. falciparum malaria among infants in a rural area of western Uganda. Participants will be recruited from four villages immediately adjacent to the Bugoye Level III Health Centre (Bugoye, Kanyanamigho, Izinga, Rwakingi 1a) in the Kasese District of western Uganda.

The first phase will consist of a series of focus group sessions with mothers of young children and their male partners to gain further insight into lesu use, to include location of purchase and frequency of washing, as well as exploring initial perceptions of insecticide-treated clothing and inform the protocols for the open-label study.

The second phase will consist of a prospective, open-label study. Twenty-five (25) mothers and their young children will be provided with insecticide-treated lesus and twenty-five (25) controls who will be provided untreated lesus. After an initial visit, bi-weekly follow up, including finger-prick blood collections will continue for a period of twelve (12) weeks.

Collected blood spots will be transported to Epicentre for real-time PCR to identify sub-microscopic parasitemia and to the French Research Institute for Development (https://en.ird.fr) in Marseille, France for quantification of the mosquito salivary antigen (gSG6-P1 peptide). Remaining samples will be stored for future analysis.

ELIGIBILITY:
Inclusion Criteria:

* Adult women (age greater or equal to 18 years) with a healthy child between the ages of 6 months to 18 months from one of four eligible villages

Exclusion Criteria:

* Mother or child with HIV (and thus taking cotrimoxazole prophylaxis)

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2019-10-28 (Actual); Primary Completion 2020-03-04 (Actual); Study Completion 2020-03-04 (Actual)

PRIMARY OUTCOMES:
Reported change in frequency of use of lesu | Baseline, 12 weeks
  Self-reported, includes discontinuation of use

SECONDARY OUTCOMES:
Incidence of symptomatic malaria episodes among children | 12 weeks
  As defined by typical symptoms including fever, malaise, and convulsions.
Incidence of P. falciparum malaria parasitemia among children | 12 weeks
  As determined by quantitative PCR
Change in mosquito salivary antigen response among children | Baseline, 12 weeks
Change in mosquito salivary antigen response among mothers | Baseline, 12 weeks
Changes in hemoglobin levels among children | Baseline, 12 weeks
Changes in hemoglobin levels among mothers | Baseline, 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ross Boyce, MD, MSc, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Bugoye Level III Health Centre, Bugoye, Kasese, Uganda

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol, ICF, CSR, Analytic Code
Time Frame: 9 to 36 months following publication
Access Criteria: The investigator who proposes to use the data has approval from an IRB, IEC, or REB, as applicable, and an executed data use/sharing agreement with UNC.

REFERENCES:
- [Derived] Boyce RM, Muhindo E, Baguma E, Muhindo R, Shem B, Francois R, Hawke S, Shook-Sa BE, Ntaro M, Nalusaji A, Nyehangane D, Reyes R, Juliano JJ, Siedner MJ, Staedke SG, Mulogo EM. Permethrin-treated baby wraps for the prevention of malaria: results of a randomized controlled pilot study in rural Uganda. Malar J. 2022 Feb 23;21(1):63. doi: 10.1186/s12936-022-04086-w. PMID 35197060